CLINICAL TRIAL: NCT01420120
Title: A Prospective Multicenter Registry to Evaluate Safety and Performance of REMEDY, Biodegradable Peripheral Stent for the Treatment of Occluded or Stenotic Superficial Femoral Arteries.
Brief Title: Remedy, Biodegradable Peripheral Stent Registry
Status: Completed | Type: Observational
Sponsor: be Medical (Industry)
Responsible Party: Joris Coteur, study coordinator, .be medical
Other Study IDs: BM-REM-03-003
Record Dates: First submitted 2011-08-16; First posted 2011-08-19 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Peripheral Arterial Disease
Keywords: Biodegradable stent, PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective multicenter registry to evaluate safety and performance of the REMEDY, biodegradable peripheral stent for the treatment of occluded or stenotic superficial femoral arteries. Patients will be followed for a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic leg ischemia requiring treatment of SFA artery or proximal popliteal artery located within the following parameters:

  * 1 cm from the femoral bifurcation in the SFA
  * 3 cm from the proximal margin of the intercondylar fossa
* Rutherford-Becker Category 2-5. In patients with bilateral lesions, the highest Rutherford Category limb should be treated. Only 1 leg can be included.
* Single lesion which can be covered by one stent.
* Target vessel reference diameter ≥ 4 mm and ≤ 6 mm (by visual estimate)
* A patent popliteal artery free from significant stenosis (>50%) with at least one patent vessel runoff as confirmed by baseline angiography
* Signed informed consent.

Exclusion Criteria:

* Pregnancy
* Previous stenting of target lesion
* Acute ischemia
* Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion). Inclusion of a patient is allowed in case inflow lesions are successfully treated during the index-procedure yielding less than 30% diameter stenosis.
* Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
* Known intolerance to study medications or contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented symptomatic occlusion and/or > 70% stenosis of SFA.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Absence of clinically driven target lesion revascularization at 12 months. | 12 months

SECONDARY OUTCOMES:
Technical success | During procedure
  Defined as a successful access and deployment of the device and determined by less than 30% residual stenosis by angiography at the baseline procedure.
Clinical success | During procedure
  Defined as technical success without the occurrence of serious adverse events during procedure
Primary and secondary patency rate | 12 months
  defined as < 50% diameter reduction and peak systolic velocity < 2.4 at 12 months.
Ankle-Brachial Index improvement of ≥ 0.1 | 1, 6 and 12 months
Clinically driven target vessel revascularization | 6 and 12 months
Major complications at 6 and 12 months, including amputation of a part of the foot, the leg below and above the knee. | 6 and 12 months
Rutherford-Becker classification of chronic limb ischemia | 1, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium